CLINICAL TRIAL: NCT01924533
Title: A Randomized, Double-blinded, Placebo Controlled, Multicentre Phase III Study to Assess the Efficacy and Safety of Olaparib (AZD2281) in Combination With Paclitaxel, Compared to Placebo in Combination With Paclitaxel, in Asian Patients With Advanced Gastric Cancer (Including the Gastro-oesophageal Junction) Who Have Progressed Following First Line Therapy
Brief Title: Efficacy and Safety Study of Olaparib in Combination With Paclitaxel to Treat Advanced Gastric Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D081BC00004
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — olaparib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaparib+ paclitaxel (Experimental): olaparib + paclitaxel
  Interventions: Drug: Olaparib; Drug: Paclitaxel
- Placebo+paclitaxel (Placebo Comparator): placebo+ paclitaxel
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Olaparib — Tablets-at a dose of 100mg orally twice daily, throughout each cycle (28 days); Once paclitaxel dosing is stopped, the planned monotherapy olaparib dose will be 300mg twice daily.
  Arms: Olaparib+ paclitaxel
Drug: Paclitaxel — IV infusion over 1 hour at 80 mg/m2 weekly on days 1, 8 and 15 of a 28 days schedule.
Drug: Placebo — Tablets-at a dose of 100mg orally twice daily, throughout each cycle (28 days); Once paclitaxel dosing is stopped, the planned monotherapy placebo dose will be 300mg twice daily.
  Arms: Placebo+paclitaxel

SUMMARY:
This study is a phase III, multi-centre study of olaparib in combination with paclitaxel, compared with placebo in combination with paclitaxel in patients with advanced gastric cancer who have progressed following first-line therapy. Patients will be from China, Japan , Korea and Taiwan.

DETAILED DESCRIPTION:
A randomized, double-blinded, multicentre phase III study to access the efficacy and safety of olaparib in combination with paclitaxel, compared with placebo in combination with paclitaxel in Asian patients with advanced gastric cancer (including gastro-oesophageal junction) who have progressed following first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced gastric cancer (including GEJ) that has progressed following first-line therapy.
* Patients must be ≥18 years of age. Age ≥20 if Japanese
* Provision of tumour sample (from either a resection or biopsy).
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed by imaging (CT/MRI) at baseline and following up visits.

Exclusion Criteria:

* More than one prior chemotherapy regimen (except for adjuvant/neoadjuvant chemotherapy with more than 6 month wash out period) for the treatment of gastric cancer in the advanced setting.
* Any previous treatment with a Polyadenosine 5'-diphosphoribose [poly-(ADP-ribose)] polymerisation (PARP) inhibitor, including olaparib.
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥5 years.
* Human Epidermalgrowth Factor Receptor-2 (HER2) positive patients.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, MD, Principal Investigator — Seoul National University, College of Medicine and Cancer Research Institute, Republic of Korea
Locations (41):
- China (17):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Ürümqi
  - Research Site, Wanzhou
  - Research Site, Wuhan
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- Japan (13):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Kasama-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Sapporo
  - Research Site, Takatsuki-shi
  - Research Site, Utsunomiya
  - Research Site, Yokohama
- South Korea (6):
  - Research Site, Anyang-si
  - Research Site, Daegu
  - Research Site, Hwasun-gun
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Taiwan (5):
  - Research Site, Kaohsiung Hsien
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bang YJ, Xu RH, Chin K, Lee KW, Park SH, Rha SY, Shen L, Qin S, Xu N, Im SA, Locker G, Rowe P, Shi X, Hodgson D, Liu YZ, Boku N. Olaparib in combination with paclitaxel in patients with advanced gastric cancer who have progressed following first-line therapy (GOLD): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Dec;18(12):1637-1651. doi: 10.1016/S1470-2045(17)30682-4. Epub 2017 Nov 2. PMID 29103871
- See also: Study protocol-redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1856&filename=GOLD%20Study%20protocol-redacted.pdf
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081BC00004&attachmentIdentifier=65ef6d55-2b26-4d0d-a8d4-d96af57903de&fileName=d081bc00004-study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants in the participant flow (525) includes all participants who were eligible and assigiend to each treatment group.
Groups:
- Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2: Olaparib 100 mg tablets bd + Paclitaxel 80 mg/m^2
- Placebo Tablets bd + Paclitaxel 80 mg/m^2: Placebo tablets bd + Paclitaxel 80 mg/m^2
Period: Overall Study
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Started | 263 | 262
Completed | 74 | 57
Not Completed | 189 | 205
Not completed — Death | 181 | 200
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Other Eligibility criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2 | Total
Number analyzed (Participants) | 263 | 262 | 525
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (11.90) [22 to 79] | 57.3 (11.14) [26 to 83] | 57.2 (11.52) [22 to 83]
Age, Continuous [Mean (Standard Deviation); unit: Years] — ATM Negative Population Population: The numbers of ATM negative population are 48 and 46 while the numbers of overall population are 263 and 262. ATM negative population is a subset of the overall population.
  Years
    number analyzed (Participants) | 48 | 46 | 94
    (all) | 57.0 (12.08) | 60.9 (9.90) | 58.9 (11.18)
Age, Customized [Count of Participants; unit: Participants]
  >=18 - <50 | 68 | 64 | 132
  >=50 - <65 | 115 | 128 | 243
  >=65 | 80 | 70 | 150
Age, Customized [Count of Participants; unit: Participants] — ATM Negative Population Population: The numbers of ATM negative population are 48 and 46 while the numbers of overall population are 263 and 262. ATM negative population is a subset of the overall population.
  Participants
    >=18 - <50: number analyzed (Participants) | 48 | 46 | 94
    >=18 - <50 | 12 | 7 | 19
    >=50 - <65: number analyzed (Participants) | 48 | 46 | 94
    >=50 - <65 | 22 | 24 | 46
    >=65: number analyzed (Participants) | 48 | 46 | 94
    >=65 | 14 | 15 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 77 | 166
  Male | 174 | 185 | 359
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic Or Latino | 263 | 262 | 525
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 263 | 262 | 525
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — ATM Negative Population Population: The numbers of ATM negative population are 48 and 46 while the numbers of overall population are 263 and 262. ATM negative population is a subset of the overall population.
  Participants
    Not Hispanic or Latino: number analyzed (Participants) | 48 | 46 | 94
    Not Hispanic or Latino | 48 | 46 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — ATM Negative Population Population: The numbers of ATM negative population are 48 and 46 while the numbers of overall population are 263 and 262. ATM negative population is a subset of the overall population.
  Participants
    Asian: number analyzed (Participants) | 48 | 46 | 94
    Asian | 48 | 46 | 94
ATM Status [Number; unit: Participants]
  Negative | 48 | 46 | 94
  Positive | 200 | 196 | 396
  Unknown | 15 | 20 | 35
Gastrectomy Status [Count of Participants; unit: Participants]
  Full | 50 | 68 | 118
  None | 136 | 122 | 258
  Partial | 77 | 72 | 149
Gastrectomy Status [Count of Participants; unit: Participants] — ATM Negative Population Population: The numbers of ATM negative population are 48 and 46 while the numbers of overall population are 263 and 262. ATM negative population is a subset of the overall population.
  Participants
    Full: number analyzed (Participants) | 48 | 46 | 94
    Full | 13 | 13 | 26
    Partial: number analyzed (Participants) | 48 | 46 | 94
    Partial | 19 | 12 | 31
    None: number analyzed (Participants) | 48 | 46 | 94
    None | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from the date of randomization until death due to any cause
Time Frame: Survival contact from the date of randomization and then every 8 weeks following objective disease progression and in the 7 days following OS Data Cut off (DCO); Time point(s) at which outcome measure is assessed up to 4 years
Population: Full analysis set population
Measure: Number; unit: participants
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 263 | 262
participants | 82 | 62
Statistical Analysis 1: Comparison: Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 vs Placebo Tablets bd + Paclitaxel 80 mg/m^2; Test type: Superiority or Other; p = 0.0262, Cox proportional hazards model; Hazard Ratio (HR) = 0.79, 97.5% CI 2-sided [0.63 to 1.00]

2. Primary Outcome: Overall Survival
Description: Time from the date of randomization until death due to any cause
Time Frame: as for outcome 1
Population: Full analysis set - ATM negative population
Measure: Number; unit: participants
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 48 | 46
participants | 19 | 11
Statistical Analysis 1: Comparison: Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 vs Placebo Tablets bd + Paclitaxel 80 mg/m^2; Test type: Superiority or Other; p = 0.2458, Cox proportional hazards model; Hazard Ratio (HR) = 0.73, 97.5% CI 2-sided [0.40 to 1.34]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time from randomization until the date of objective radiological disease progression according to RECIST (v1.1) or death by any cause in the absence of progression. Objective progression is defined as at least a 20% increase in the sum of the diameters of the target lesions (compared to previous minimum sum) or an overall non-target lesion assessment of progression or a new lesion.
Time Frame: Scans taken at baseline and then follow up assessments taken every 8 weeks up to Week 40 and then every 16 weeks until objective disease progression as defined by RECIST 1.1, assessed up to 3 years
Population: FAS analysis set population
Measure: Number; unit: participants
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 263 | 262
participants | 47 | 29
Statistical Analysis 1: Comparison: Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 vs Placebo Tablets bd + Paclitaxel 80 mg/m^2; Test type: Superiority or Other; p = 0.0645, Cox proportional hazards model; Hazard Ratio (HR) = 0.84, 97.5% CI 2-sided [0.67 to 1.04]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: FAS analysis set - ATM negative population
Measure: Number; unit: participants
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 48 | 46
participants | 11 | 7
Statistical Analysis 1: Comparison: Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 vs Placebo Tablets bd + Paclitaxel 80 mg/m^2; Test type: Superiority or Other; p = 0.2199, Cox proportional hazards model; Hazard Ratio (HR) = 0.74, 97.5% CI 2-sided [0.42 to 1.29]

5. Secondary Outcome: Number of Patients With Objective Response.
Description: Number of patients with objective response. Per RECIST 1.1, complete response (CR) is disappearance of all target lesions since baseline; partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions. Overall Response = CR + PR.
Time Frame: as for outcome 3
Population: Full analysis set population
Measure: Number; unit: participants
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 263 | 262
participants | 44 | 28
Statistical Analysis 1: Comparison: Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 vs Placebo Tablets bd + Paclitaxel 80 mg/m^2; Test type: Superiority or Other; p = 0.0548, Regression, Logistic; Odds Ratio (OR) = 1.69, 97.5% CI 2-sided [0.92 to 3.17]

6. Secondary Outcome: Number of Patients Objective Response
Description: as for outcome 5
Time Frame: as for outcome 3
Population: Full analysis set - ATM negative population
Measure: Number; unit: participants
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 48 | 46
participants | 12 | 5
Statistical Analysis 1: Comparison: Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 vs Placebo Tablets bd + Paclitaxel 80 mg/m^2; Test type: Superiority or Other; p = 0.0309, Regression, Logistic; Odds Ratio (OR) = 4.24, 97.5% CI 2-sided [0.95 to 23.23]

7. Secondary Outcome: Number of Patients With Deterioration of Health Related Quality of Life (HRQoL) as Assessed by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Questionnaire Core 30 Item Module (QLQ-C30) Global HRQoL Scale
Description: Number of patients with a clinically important deterioration in the global HRQoL score or death by any cause in the absence of a clincially meaningful symptom deterioration
Time Frame: Pre-treatment , Day 29 and then every 4 weeks until discontinuation, assessed up to 3 years
Population: Patients whose baseline HRQoL score >=10 in full analysis set population
Measure: Number; unit: participants
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 240 | 249
participants | 160 | 177
Statistical Analysis 1: Comparison: Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 vs Placebo Tablets bd + Paclitaxel 80 mg/m^2; Test type: Superiority or Other; p = 0.0716, Cox proportional hazards model; Hazard Ratio (HR) = 0.82, 97.5% CI 2-sided [0.64 to 1.05]

8. Secondary Outcome: Number of Patients With Deterioration of Health Related Quality of Life (HRQoL) as Assessed by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Questionnaire Core 30 Item Module (QLQ-C30) Global HRQoL Scale
Description: as for outcome 7
Time Frame: Pre-treatment , Day 29 and then every 4 weeks until discontinuation, assessed up to 3 years
Population: Patients whose baseline HRQoL score >=10 in full analysis set ATM negative population
Measure: Number; unit: participants
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 41 | 43
participants | 29 | 33
Statistical Analysis 1: Comparison: Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 vs Placebo Tablets bd + Paclitaxel 80 mg/m^2; Test type: Superiority or Other; p = 0.0927, Cox proportional hazards model; Hazard Ratio (HR) = 0.63, 97.5% CI 2-sided [0.34 to 1.16]

9. Secondary Outcome: Time to Response
Description: Time from randomization to the first onset of a confirmed objective tumour response
Time Frame: as for outcome 3
Population: Patients with objective response in full analysis set population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 44 | 28
days | 57.0 [54.5 to 64.0] | 57.0 [56.0 to 111.5]

10. Secondary Outcome: Time to Response
Description: Time from randomization to the first onset of a confirmed objective tumour response
Time Frame: as for outcome 3
Population: Patients with objective response in full analysis set ATM negative population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 12 | 5
days | 57.5 [57.0 to 113.0] | 57.0 [55.0 to 58.0]

11. Secondary Outcome: Duration of Response
Description: Time from the first documentation of CR/PR until the date of progression, or the last evaluable RECIST assessment for patients taht do not progress or progress after two or more missed visits
Time Frame: as for outcome 3
Population: Patients with objective response in full analysis set population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 44 | 28
days | 166.0 [89.0 to 218.0] | 64.0 [54.0 to 186.0]

12. Secondary Outcome: Duration of Response
Description: as for outcome 11
Time Frame: as for outcome 3
Population: Patients with objective response in full analysis set ATM negative population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 12 | 5
days | 171.0 [124.0 to 350.0] | 108.0 [57.0 to 113.0]

ADVERSE EVENTS:
Description: Participants in the Full Analysis Set (i.e., 263 and 262) were monitored/assessed for All-Cause Mortality/Overall Survival and participants in the Safety Set (i.e., 262 and 259) were monitored/assessed for Serious and Other (Not Including Serious) Adverse Events.
Arm/Group | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 | Placebo Tablets bd + Paclitaxel 80 mg/m^2
All-Cause Mortality (participants affected / at risk) | 181/263 | 200/262
Serious Adverse Events (participants affected / at risk) | 92/262 | 65/259
Other Adverse Events (participants affected / at risk) | 257/262 | 253/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 (N=262) | Placebo Tablets bd + Paclitaxel 80 mg/m^2 (N=259)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Bone marrow disorder (Blood and lymphatic system disorders) | 6 (7) | 3 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Granulocytopenia (Blood and lymphatic system disorders) | 5 (6) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4) | 4 (5)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 1 (2)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4)
Asthenia (General disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 4 (5) | 4 (4)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 3 (3) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 4 (4)
Scrub typhus (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Coagulation test abnormal (Investigations) | 1 (1) | 0 (0)
Granulocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Stent malfunction (Product Issues) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Venous thrombosis (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 100 mg Tablets bd + Paclitaxel 80 mg/m^2 (N=262) | Placebo Tablets bd + Paclitaxel 80 mg/m^2 (N=259)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (21) | 15 (26)
Anaemia (Blood and lymphatic system disorders) | 99 (156) | 62 (101)
Leukopenia (Blood and lymphatic system disorders) | 71 (232) | 57 (177)
Neutropenia (Blood and lymphatic system disorders) | 122 (373) | 108 (300)
Abdominal distension (Gastrointestinal disorders) | 19 (22) | 19 (20)
Abdominal pain (Gastrointestinal disorders) | 23 (26) | 28 (33)
Abdominal pain upper (Gastrointestinal disorders) | 20 (23) | 15 (17)
Constipation (Gastrointestinal disorders) | 38 (52) | 50 (63)
Diarrhoea (Gastrointestinal disorders) | 66 (102) | 51 (65)
Dyspepsia (Gastrointestinal disorders) | 13 (14) | 13 (16)
Nausea (Gastrointestinal disorders) | 75 (121) | 63 (93)
Stomatitis (Gastrointestinal disorders) | 21 (32) | 12 (13)
Vomiting (Gastrointestinal disorders) | 45 (67) | 43 (70)
Asthenia (General disorders) | 45 (50) | 35 (51)
Fatigue (General disorders) | 48 (70) | 52 (71)
Malaise (General disorders) | 15 (41) | 12 (23)
Pyrexia (General disorders) | 34 (45) | 36 (59)
Nasopharyngitis (Infections and infestations) | 16 (20) | 9 (16)
Upper respiratory tract infection (Infections and infestations) | 19 (31) | 14 (16)
Alanine aminotransferase increased (Investigations) | 31 (40) | 14 (18)
Aspartate aminotransferase increased (Investigations) | 23 (27) | 16 (22)
Blood bilirubin increased (Investigations) | 10 (13) | 14 (15)
Haemoglobin decreased (Investigations) | 18 (35) | 20 (37)
Neutrophil count decreased (Investigations) | 67 (188) | 38 (80)
Platelet count decreased (Investigations) | 20 (28) | 12 (18)
White blood cell count decreased (Investigations) | 60 (165) | 48 (116)
Decreased appetite (Metabolism and nutrition disorders) | 86 (127) | 69 (97)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 (16) | 13 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 21 (25) | 16 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 13 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 37 (51) | 35 (65)
Dizziness (Nervous system disorders) | 11 (14) | 14 (14)
Hypoaesthesia (Nervous system disorders) | 20 (23) | 16 (18)
Neuropathy peripheral (Nervous system disorders) | 41 (41) | 42 (45)
Peripheral sensory neuropathy (Nervous system disorders) | 41 (45) | 29 (30)
Insomnia (Psychiatric disorders) | 20 (22) | 19 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (29) | 24 (27)
Alopecia (Skin and subcutaneous tissue disorders) | 112 (112) | 116 (117)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (13) | 17 (18)
Rash (Skin and subcutaneous tissue disorders) | 35 (44) | 24 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 60 days prior to submission of any material for publication or presentation, Institution and Principal Investigator (PI) shall jointly provide AstraZeneca with such material for review. If requested in writing by AstraZeneca, Institution and PI shall withhold material from submission for publication or presentation for an additional 90 days from the date of AstraZeneca's request to allow for the filing patent application or preserve its proprietary rights in the information.